CLINICAL TRIAL: NCT06794528
Title: A Randomized Two-Arm Clinical Trial, Fixed-Assignment Study on Adherence to Therapeutic Exercise in Cervical Rehabilitation Using A Serious Game In Mobile Devices
Brief Title: Therapeutic Exercise Through Exergames on Mobile Devices for Cervical Rehabilitation
Acronym: RehbeCa
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat de les Illes Balears (Other)
Responsible Party: Principal Investigator, Iosune Salinas-Bueno, Principal Investigator, Universitat de les Illes Balears
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TED2021-131358A-I00_RCT; TED2021-131358A-I00 (Other Grant/Funding Number: Granted by MICIU/AEI/10.13039/501100011033)
Record Dates: First submitted 2025-01-20; First posted 2025-01-27 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Home exercise via mobile App (Experimental): During two months, participants will be asked to use the therapeutic exercise game in the application three times a week.
  Interventions: Other: RehbeCa mobile application
- Usual home exercise program (Active Comparator): During two months, participants will be asked to performed the therapeutic exercise, previously explained, three times a week.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: RehbeCa mobile application — The system consists of a mobile application (to be used by patients) and a web application (to be used by physiotherapists) that allows monitoring of the patient's performance without the need for attendance, thus facilitating telerehabilitation. The mobile application consists of a serious game that aims to induce the patient to perform neck exercises, adapting to their capacity and evolution at all times through artificial intelligence. The patient's interaction with the mobile application is based on the integration of a vision-based head-tracker to track the movements of the patient's head. The web application aims to provide professionals with a tool to monitor the evolution of their patients through the data captured by the mobile application.
  Other Names: RehbeCa application system
  Arms: Home exercise via mobile App
Other: Home exercise program — Set of therapeutic exercises to be carried out at home. They are taught face-to-face, and also printed on a leaflet that is delivered to the participant.
  Arms: Usual home exercise program

SUMMARY:
The objective of this study is to determine whether performing cervical therapeutic exercises using a serious game through a mobile application enhances treatment adherence compared to performing the same exercises at home following standard practice.

DETAILED DESCRIPTION:
Participants in the study will be adults with non-specific neck pain (cervicalgia) who own a smartphone or tablet, and that give informed consent. Individuals with acute or severe conditions, such as recent surgeries or trauma, will be excluded. Before participation, they will be informed about the study and potential risks. The study is designed as a randomized clinical trial with two groups. The control group will follow a traditional home exercise program with written instructions, while the intervention group will use a personalized mobile app to guide their exercises. All participants will be asked to log their progress and any incidents in a compliance journal.

ELIGIBILITY:
Inclusion Criteria:

* Persons of legal age with cervicalgia.
* Have a smart mobile device (smartphone or tablet) on which to download the App.

Exclusion Criteria:

* Acute musculoskeletal pathological processes or exacerbation (less than 15 days of evolution). Includes presentation of symptoms such as paraesthesia, radiating pain, loss of strength in the upper limb.
* Episodes of severe pain more than 15 days of evolution.
* Accident with cervical or dorsal injury within the last month.
* Refusing to sign the informed consent.
* Not having a device suitable for installation or lack of experience in the use of smart mobile devices.
* Baseline NDI score of less than 5.
* Presence of red flags:

  * Suspicion of fracture: advanced age, previous trauma, osteoporosis.
  * Suspicion of neurological involvement: loss of sensation in extremities, loss of strength or muscle mass.
  * Suspicion of infection: fever, night sweats.
  * Suspicion of cancer: Previous history of cancer, no improvement in one month of treatment, weight loss, headache, vomiting.
  * Suspicion of systemic disease: headache, fever, malaise, general headache, fever, malaise, unilateral skin rash (herpes).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-16 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Level of Compliance of the Exercise Prescription | From admission to discharge, every 15 days, up to two months.
  The level of compliance is a percentage showing the difference between the self-reported performed sessions, reflected in the compliance diary, and the prescribed sessions.Possible score ranges from 0% to 100%, considering compliant participants over 80%.

SECONDARY OUTCOMES:
Changes in Pain Intensity | Baseline and every 15 days, up to two months.
  Pain intensity measured with Visual Analogue Scale (VAS). Possible scores range from 0 (no pain) to 10 (worst possible pain).
Changes in Neck disability | Baseline and every 15 days, up to two months.
  Level of disability caused by neck pain, measured by Neck Disability Index (NDI) questionnaire. NDI is widely used to evaluate the impact of neck pain on daily activities. It is a questionnaire with 10 items about pain, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation. Item responses range from 0 (no pain) to 5 (worst imaginable pain). The 10 responses are summed to a score from 0 to 50 with higher scores indicating more disability. The NDI categories are no disability (0-4 points), mild disability (5-14 points), moderate disability (15-24 points), severe disability (25-34 points) or complete disability (35-50 points)
Changes in Cervical Active Range of Motion | Baseline and every 15 days, up to two months.
  Active Range of Motion (ROM) of the neck, measured recording real-time movements with validated ENLAZA inertial sensors (Werium Assistive Solutions S.L., 2022). ROM measurements collected will be flexion (0-45º), extension (0-45º), lateral flexion (0-45º each side), and neck rotation (0-70º each side).

CONTACTS AND LOCATIONS:
Locations (1):
- University of the Balearic Islands, Palma de Mallorca, Balearic Islands, Spain

IPD SHARING:
Plan to Share IPD: Yes
Socio-demographic data and health data such as pain scores, ROM records or adherence to treatment will be collected deidentified. All data will be recorded in the data processing register RAT Code 034 of the University of the Balearic Islands: 'Therapeutic Exercise Through Exergames on Mobile Devices or Cervical Rehabilitation" All the individual data collected during the trial will be shared, after deidentification. Also, study protocol will be available. Dataset will be available following publication of results, for any purposes, at Institutional Data Repository CORA. RDR, a federated data repository that allows publishing datasets in a FAIR way and following the guidelines of the European Open Science Cloud (EOSC).
Supporting Information: Study Protocol
Time Frame: Following publication of results, no end date.
Access Criteria: Available

REFERENCES:
- [Background] Jahre H, Grotle M, Smedbraten K, Dunn KM, Oiestad BE. Risk factors for non-specific neck pain in young adults. A systematic review. BMC Musculoskelet Disord. 2020 Jun 9;21(1):366. doi: 10.1186/s12891-020-03379-y. PMID 32517732
- [Background] Cheng CH, Su HT, Yen LW, Liu WY, Cheng HY. Long-term effects of therapeutic exercise on nonspecific chronic neck pain: a literature review. J Phys Ther Sci. 2015 Apr;27(4):1271-6. doi: 10.1589/jpts.27.1271. Epub 2015 Apr 30. PMID 25995604
- [Background] Zronek M, Sanker H, Newcomb J, Donaldson M. The influence of home exercise programs for patients with non-specific or specific neck pain: a systematic review of the literature. J Man Manip Ther. 2016 May;24(2):62-73. doi: 10.1179/2042618613Y.0000000047. PMID 27559275
- [Background] Minghelli B. Musculoskeletal spine pain in adolescents: Epidemiology of non-specific neck and low back pain and risk factors. J Orthop Sci. 2020 Sep;25(5):776-780. doi: 10.1016/j.jos.2019.10.008. Epub 2019 Nov 7. PMID 31708228
- [Background] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503
- [Background] Noormohammadpour P, Tayyebi F, Mansournia MA, Sharafi E, Kordi R. A concise rehabilitation protocol for sub-acute and chronic non-specific neck pain. J Bodyw Mov Ther. 2017 Jul;21(3):472-480. doi: 10.1016/j.jbmt.2016.07.005. Epub 2016 Jul 25. PMID 28750953
- [Background] Bailey DL, Holden MA, Foster NE, Quicke JG, Haywood KL, Bishop A. Defining adherence to therapeutic exercise for musculoskeletal pain: a systematic review. Br J Sports Med. 2020 Mar;54(6):326-331. doi: 10.1136/bjsports-2017-098742. Epub 2018 Jun 6. PMID 29875278
- [Background] Ayed I, Ghazel A, Jaume-I-Capo A, Moya-Alcover G, Varona J, Martinez-Bueso P. Vision-based serious games and virtual reality systems for motor rehabilitation: A review geared toward a research methodology. Int J Med Inform. 2019 Nov;131:103909. doi: 10.1016/j.ijmedinf.2019.06.016. Epub 2019 Jul 10. PMID 31557701
- [Background] Manresa-Yee, C., Ponsa, P., Salinas, I., Perales, F.J., Negre, F., Varona, J. (2014). Observing the use of an input device for rehabilitation purposes. Behav. Inf. Technol. 33, 3, 271-282.
- [Background] Roig-Maimo MF, Manresa-Yee C, Varona J. A Robust Camera-Based Interface for Mobile Entertainment. Sensors (Basel). 2016 Feb 19;16(2):254. doi: 10.3390/s16020254. PMID 26907288
- [Background] Ayed I, Ghazel A, Jaume-I-Capo A, Moya-Alcover G, Varona J, Martinez-Bueso P. Feasibility of Kinect-Based Games for Balance Rehabilitation: A Case Study. J Healthc Eng. 2018 Jul 9;2018:7574860. doi: 10.1155/2018/7574860. eCollection 2018. PMID 30123443
- [Background] Salinas-Bueno I, Roig-Maimo MF, Martinez-Bueso P, San-Sebastian-Fernandez K, Varona J, Mas-Sanso R. Camera-Based Monitoring of Neck Movements for Cervical Rehabilitation Mobile Applications. Sensors (Basel). 2021 Mar 23;21(6):2237. doi: 10.3390/s21062237. PMID 33806813